CLINICAL TRIAL: NCT02577835
Title: International Registry for Ambulatory Blood Pressure and Arterial Stiffness Telemonitoring
Acronym: VASOTENS
Status: Completed | Type: Observational
Sponsor: Italian Institute of Telemedicine (Other)
Collaborators: BPLab (Other)
Responsible Party: Sponsor
Other Study IDs: VASOTENS REGISTRY
Record Dates: First submitted 2015-10-13; First posted 2015-10-16 (Estimated); Results first posted 2024-03-01 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: Hypertension
Keywords: Hypertension; Arterial Stiffness; Ambulatory blood pressure
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypertensive patients: No intervention. Patients will be sumbitted to standard tests required for hypertension management, including ambulatory blood pressure monitoring, and pharmacologically treated according to recommendations of international guidelines. The registry will include data from subjects fulfilling the inclusion criteria and whose data are contained in existing databases collected by the participating centers and who are regularly followed-up at the center. New subjects can be enrolled for this project, but they must be submitted to ambualtory blood pressure monitoring because it is required for evaluating their hypertension status, according to current recommendations.
  Interventions: Device: Ambulatory blood pressure monitoring

INTERVENTIONS:
Device: Ambulatory blood pressure monitoring — Ambulatory blood pressure monitoring with arterial stiffness evaluation at 6-12 month intervals.

SUMMARY:
This Registry is an investigator-initiated, international, multicenter, observational, prospective study aiming at: i) evaluating non-invasive 24-h ambulatory blood pressure and arterial stiffness estimates (through 24-h pulse wave analysis) in hypertensive subjects; ii) assessing the changes in estimates following treatment; iii) weighing the impact of 24-h pulse wave analysis on target organ damage and cardiovascular prognosis; iv) assessing the relationship between arterial stiffness, blood pressure absolute level and variability, and prognosis. Approximately 2000 subjects, referred to 20 hypertension clinics for routine diagnostic evaluation and follow-up of hypertension, will be recruited. Data collection will include ambulatory blood pressure monitoring, performed with a device allowing simultaneous non-invasive assessment of blood pressure and arterial stiffness, and clinical data (including cardiovascular outcomes). A web-based telemedicine platform will be used for data collection. Subjects will visit the centers at 6-12 month intervals. First follow-up results are expected to be available in the next 2-years. The results of the Registry will help defining the normalcy thresholds for current and future indices derived from 24-h pulse wave velocity, according to outcome data. They will also provide supporting evidence for the inclusion of such evaluation in recommendations on hypertension management.

DETAILED DESCRIPTION:
The VASOTENS Registry is an international, multicenter, observational, prospective project Actually, it is a large database of ambulatory blood pressure recordings obtained with a non-invasive device, able to determine central blood pressure and various indices of arterial stiffness (mainly pulse wave velocity and augmentation index) over the 24-hours, based on a clinically validated technology of pulse wave analysis of oscillometric blood pressure measurements, integrated in an ambulatory blood pressure monitor. Specifically, this project aims at creating an international network of centers performing ambulatory blood pressure monitoring and arterial stiffness monitoring, in order to evaluate the impact of such estimates on the clinical outcome of hypertensive patients. The results of the data collected at baseline and during regular follow-up of hypertensive patients (up to 2 years) will help to provide evidence on the clinical usefulness of such technologies for the screening and follow-up of the hypertensive patients. The registry will include data from subjects fulfilling the inclusion criteria and whose data are contained in existing databases collected by the participating centers and who are regularly followed-up at the center. New subjects can be enrolled for this project, but they must be submitted to ambulatory blood pressure monitoring because it is required for evaluating their hypertension status, according to current recommendations. Data collection is ensured by a dedicated web-based telemedicine platform, including an electronic case report form (e-CRF). The e-CRF allows collection of patient's clinical data, such as family history, anthropometric data, habits, past and current diseases, therapies, office blood pressure, and laboratory tests, including evaluation of target organ damage. The project does not involve any type of intervention related to the study and the physicians can manage the patients included in the Registry according to the requirements of clinical practice and current guidelines. However, as recommended by current guidelines, each patient has to be followed-up with visits occurring at regular intervals (ideally every 6 months, and not less than once a year). The physicians is also free to use the ambulatory blood pressure data in the clinical management of the patients. At least 30 Hypertension centers are planned to be involved in the project, each one providing at least 100 patients, which have to be followed-up over time. Centers will be selected in different countries, initially in Europe, starting from Italy and Russia. Mandatory criteria of a center to be included in the study are the availability in the facility of a BPLab ambulatory blood pressure monitor, the potential for providing and properly following-up the number of patients required by the protocol, the availability of Internet connection, regular access to the web and human resources to upload ambulatory blood pressure and clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Subjects referred to routine diagnostic evaluation for hypertension or established hypertensive subject
* ABPM performed for clinical reasons with a BPLab device
* Valid ambualtory blood pressure recordings (interval between measurements not >30 minutes, at least 70% of expected number of readings, at least 20 valid readings during the day-time and 7 during the night-time)
* Availability of individual measurements for ambulatory blood pressure monitoring
* Availability of basic demographic and clinical information
* Availability of a signed informed consent form

Exclusion Criteria:

* Age <18 years
* Atrial fibrillation, frequent ectopic beats, second or third degree atrioventricular blocks, or other conditions which might make difficult or unreliable the automatic blood pressure measurement with the oscillometric technique
* Upper arm circumference <22 cm
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected hypertensive patients referred to routine diagnostic evaluation for their condition (hypertension) or established hypertensive subjects
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2022-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Omboni, MD, Study Chair — Italian Institute of Telemedicine
Locations (24):
- Argentina (2):
  - DIM Clinica Privada, Buenos Aires
  - Servicio de Clínica Médica y Sección Hipertensión Arterial, Hospital Italiano de Buenos Aires, Buenos Aires
- Center of Preventive Cardiology, Yerevan, Armenia
- Department of Biomedical Sciences, Faculty of Medicine and Health Sciences, Macquarie University, Sydney, Australia
- Italy (2):
  - Dipartimento di Scienze Mediche e Chirurgiche, Università di Brescia, Medicina 2, Spedali Civili, Brescia
  - Unità Operativa di Nefrologia ed Ipertensione, Centro di Riferimento Regionale per l'Ipertensione Arteriosa, Policlinico Paolo Giaccone, Palermo
- Department of Functional Diagnostics, Medical Centre Hospital of President's Affairs Administration of The Republic of Kazakhstan, Astana, Kazakhstan
- University of Guadalajara, Dept. of Physiology, Guadalajara, Mexico
- Portugal (2):
  - Clínica da Aveleira, Instituto de Investigação e Formação Cardiovascular, Coimbra
  - Escola Superior de Tecnologia da Saúde de Coimbra , Instituto Politécnico de Coimbra, Coimbra
- Cardiac Rehabilitation Clinic, Tirgu Mures Emergency Clinical County Hospital, Târgu Mureş, Romania
- Russia (12):
  - South Ural State Medical University, Chelyabinsk
  - Diagnostics Department, The Hospital within the Russian Railroad Network, Chita
  - Department of Cardiology and Personalized Medicine, Faculty of Doctors' Advanced Training, Peoples' Friendship University of Russia, Moscow
  - Department of Cardiology, Sechenov First Moscow State Medical University, Moscow
  - Department of Propaedeutics of Internal Diseases, Medical Faculty, Peoples' Friendship University of Russia, Moscow
  - Institute of Personalized Medicine, Sechenov First Moscow State Medical University, Moscow
  - Lomonosov Moscow State University Clinic, State University, Moscow
  - Volga District Medical Center, Nizhny Novgorod
  - Petrosavodsk Research Center and Department of Faculty Therapy, Infectious Diseases and Epidemiology, Petrozavodsk State University, Petrozavodsk
  - Rostov State Medical University, Rostov-at-Don
  - North-West Federal Medical Research Centre, Department of Epidemiology, Saint Petersburg
  - Volgograd State Medical University, Volgograd
- National Scientific Center "M.D. Strazhesko Institute of Cardiology", Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Omboni S, Posokhov IN, Parati G, Avolio A, Rogoza AN, Kotovskaya YV, Mule G, Muiesan ML, Orlova IA, Grigoricheva EA, Cardona Munoz E, Zelveian PH, Pereira T, Peixoto Maldonado JM. Vascular Health Assessment of The Hypertensive Patients (VASOTENS) Registry: Study Protocol of an International, Web-Based Telemonitoring Registry for Ambulatory Blood Pressure and Arterial Stiffness. JMIR Res Protoc. 2016 Jun 29;5(2):e137. doi: 10.2196/resprot.5619. PMID 27358088
- [Background] Omboni S, Posokhov IN, Kotovskaya YV, Protogerou AD, Blacher J. Twenty-Four-Hour Ambulatory Pulse Wave Analysis in Hypertension Management: Current Evidence and Perspectives. Curr Hypertens Rep. 2016 Oct;18(10):72. doi: 10.1007/s11906-016-0681-2. PMID 27659178
- [Background] Omboni S, Campolo L, Panzeri E. Telehealth in chronic disease management and the role of the Internet-of-Medical-Things: the Tholomeus(R) experience. Expert Rev Med Devices. 2020 Jul;17(7):659-670. doi: 10.1080/17434440.2020.1782734. Epub 2020 Jun 30. PMID 32536214
- [Background] Omboni S, Panzeri E, Campolo L. E-Health in Hypertension Management: an Insight into the Current and Future Role of Blood Pressure Telemonitoring. Curr Hypertens Rep. 2020 Jun 6;22(6):42. doi: 10.1007/s11906-020-01056-y. PMID 32506273
- [Background] Omboni S, Arystan A, Benczur B. Ambulatory monitoring of central arterial pressure, wave reflections, and arterial stiffness in patients at cardiovascular risk. J Hum Hypertens. 2022 Apr;36(4):352-363. doi: 10.1038/s41371-021-00606-4. Epub 2021 Sep 13. PMID 34518619
- [Result] Omboni S, Posokhov I, Parati G, Rogoza A, Kotovskaya Y, Arystan A, Avolio A, Barkan V, Bulanova N, Cardona Munoz E, Grigoricheva E, Konradi A, Minyukhina I, Muiesan ML, Mule G, Orlova I, Pereira T, Peixoto Maldonado JM, Statsenko ME, Tilea I, Waisman G; VASOTENS Registry Study Group. Ambulatory blood pressure and arterial stiffness web-based telemonitoring in patients at cardiovascular risk. First results of the VASOTENS (Vascular health ASsessment Of The hypertENSive patients) Registry. J Clin Hypertens (Greenwich). 2019 Aug;21(8):1155-1168. doi: 10.1111/jch.13623. Epub 2019 Jul 11. PMID 31294910
- [Result] Omboni S, Posokhov I, Parati G, Arystan A, Tan I, Barkan V, Bulanova N, Derevyanchenko M, Grigoricheva E, Minyukhina I, Mule G, Orlova I, Paini A, Peixoto Maldonado JM, Pereira T, Ramos-Becerra CG, Tilea I, Waisman G; VASOTENS Registry Study Group. Variable association of 24-h peripheral and central hemodynamics and stiffness with hypertension-mediated organ damage: the VASOTENS Registry. J Hypertens. 2020 Apr;38(4):701-715. doi: 10.1097/HJH.0000000000002312. PMID 31834122
- [Result] Omboni S, Alfie J, Arystan A, Avolio A, Barin E, Bokusheva J, Bulanova N, Butlin M, Cuffaro P, Derevyanchenko M, Grigoricheva E, Gurevich A, Konradi A, Muiesan ML, Paini A, Pereira T, Statsenko ME, Tan I; VASOTENS Registry Study Group. Association of 24-h central hemodynamics and stiffness with cardiovascular events and all-cause mortality. The VASOTENS Registry. J Hypertens. 2024 Sep 1;42(9):1590-1597. doi: 10.1097/HJH.0000000000003763. Epub 2024 May 15. PMID 38747378
- See also: The official website of the study — http://www.vasotens.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hypertensive Patients
Started | 1342
Completed | 1200
Not Completed | 142
Not completed — Ambulatory blood pressure recordings were not valid for the analysis | 142

BASELINE CHARACTERISTICS:
Arm/Group | Hypertensive Patients
Number analyzed (Participants) | 1200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 905
  >=65 years | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 536
  Male | 664
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 59
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 84
  White | 1057
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 82
  Romania | 53
  Italy | 321
  Mexico | 71
  Australia | 108
  Kazakhstan | 22
  Portugal | 144
  Russia | 399

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Pulse Wave Velocity (PWV)
Description: 24-hour average value for arterial stiffness was assessed through estimation of the time traveled by the pulse wave from the central arterial tree (aorta) to the peripheral arteries (brachial artery) and measured in meters per sec. The faster the wave travels through the arterial tree, the stiffer the artery is.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Hypertensive Patients
Number analyzed (Participants) | 1200
m/s | 10.6 (2.6)

2. Primary Outcome: 24-hour Augmentation Index (AI)
Description: 24-hour average value for waves reflection expressed as a percentage. The augmentation index is a measure of wave reflection and arterial stiffness and is commonly measured as the ratio of the central pulse pressure and the reflected pulse pressure which augments the central blood pressure. When arteries are stiff, a reflected wave is formed where arteries split. This reflected wave moves back at the heart and increases the pressure at which the heart has to pump. The higher the index the stiffer the artery is.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Hypertensive Patients
Number analyzed (Participants) | 1200
percent | 18.0 (18.6)

3. Primary Outcome: 24-hour Central Blood Pressure
Description: 24-hour average central aortic pressure expressed in mmHg, as the estimated blood pressure at the level of the thoracic aorta
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hypertensive Patients
Number analyzed (Participants) | 1200
mmHg | 117.2 (12.8)

4. Secondary Outcome: 24-hour Systolic Blood Pressure
Description: Average 24-hour brachial systolic blood pressure (mmHg), namely the systolic blood pressure measured at the level of the brachial artery (upper arm).
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hypertensive Patients
Number analyzed (Participants) | 1200
mmHg | 128.1 (14.3)

5. Secondary Outcome: 24-hour Diastolic Blood Pressure
Description: Average 24-hour brachial diastolic blood pressure (mmHg), namely the diastolic blood pressure measured at the level of the brachial artery (upper arm).
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hypertensive Patients
Number analyzed (Participants) | 1200
mmHg | 79.4 (9.6)

6. Secondary Outcome: Cardiac Damage (Left Ventricular Hypertrophy at Echocardiogram or ECG)
Description: Left ventricular mass indexed by body surface area (g/m^2) is used to identify left ventricular hypertrophy in case it is increased above a certain threshold (see protocol).
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Hypertensive Patients
Number analyzed (Participants) | 1200
g/m^2 | 109.6 (21.3)

7. Secondary Outcome: Vascular Damage (Carotid Plaque at Ultrasonography)
Description: Intima media tickness (mm) measured by carotid ultrasonography is used to identify wall thickening or atherosclerotic plaque, when it is above a certain threshold (see protocol).
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Hypertensive Patients
Number analyzed (Participants) | 1200
mm | 1.2 (0.5)

8. Secondary Outcome: Renal Damage (Urine Protein)
Description: Urine proteine (mg/24h). The increase above a certain threshold of urine protein is a sign of renal damage (see protocol).
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mg/24h
Arm/Group | Hypertensive Patients
Number analyzed (Participants) | 1200
mg/24h | 105.4 (129.2)

9. Secondary Outcome: Combination of Non-fatal and Fatal CV and Renal Events or All-cause Death
Description: The outcome variables consisted of a combination of nonfatal (i.e., not causing death) and fatal events (i.e., causing death) and all-cause death. The outcome variables included transient ischemic attack (TIA) or stroke (ischemic or hemorrhagic), myocardial infarction, angina pectoris or coronary revascularization, heart failure, peripheral vascular disease, and renal failure.
  All outcomes were recorded by the Investigator on the date of the first occurrence or on the last study visit.
Time Frame: 4 years
Population: The subgroup of patients followed for the occurrence of major cardiovascular event and all-cause death
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertensive Patients
Number analyzed (Participants) | 591
Participants | 104

ADVERSE EVENTS:
Time Frame: 4.2 years
Description: The following adverse events were collected:
  1. All-Cause Mortality: the occurrence of death due to any cause (cardiovascular and non cardiovascular)
  2. Serious Adverse Events: included nonfatal events (hospitalization) due to transient ischemic attack or stroke (ischemic or hemorragic), myocardial infarction, angina pectoris, or coronary revascularization, heart failure, peripheral vascular disease, renal failure.
  3. Other Adverse Events: not applicable for this study
Arm/Group | Hypertensive Patients
All-Cause Mortality (participants affected / at risk) | 24/591
Serious Adverse Events (participants affected / at risk) | 80/591
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypertensive Patients (N=591)
Transient Ischemic Attack (TIA) or stroke (ischemic or hemorragic) (Vascular disorders) | 24 (42)
Myocardial infarction, angina pectoris, or coronary revascularization (Cardiac disorders) | 19 (19)
Heart failure (Cardiac disorders) | 17 (17)
Peripheral vascular disease (Vascular disorders) | 7 (7)
Renal failure (Renal and urinary disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2015-02-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT02577835/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT02577835/SAP_001.pdf
  • Informed Consent Form (2015-01-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT02577835/ICF_002.pdf